CLINICAL TRIAL: NCT05636956
Title: The Effect of Education and Counseling Program on Patients With Cardiac Implantable Electronic Devices and Low Health Literacy
Brief Title: Education and Counseling Program on Patients With CIEDs and Low HL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Merve Erunal, Research Assistant, MSc., PhD(c)., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/16-34
Record Dates: First submitted 2022-11-16; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Arrhythmias, Cardiac; Heart Failure; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Failure; Behavior | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who receive education and counseling program (Experimental): Patients with CIEDs and low health literacy received education and counseling program by researchers.
  Interventions: Other: Education and Counseling Program
- Patients who receive clinical routine care (No Intervention): Patients with CIEDs and low health literacy received only clinical routine care.

INTERVENTIONS:
Other: Education and Counseling Program — Researches created an education and counseling program. In this context, patients receive an one hour education. Education program consist of face-to-face informing and teach-back method. At the end of the face-to-face informing, researchers give a comicbook about instructions of living with CIEDs as a written material. After discharge, researches follow-up patients with phone calls. In the context of phone calls researches continue to informing patients, remind related instructions for that time and answer questions of patients. Patients are allowed to reach reserarches any time if they have any concern or question. This program lasts for six months.
  Other Names: Education and counseling program about living with CIEDs.
  Arms: Patients who receive education and counseling program

SUMMARY:
The goal of this RCT (randomized controlled trial) is to investigate the effect of education and counseling program that researches developed on patients with cardiac implantable electronic devices (CIEDs) and low health literacy.

The main questions are; Is there a difference between the health literacy scores of intervention and control groups after education and counseling program? Is there a difference between the CIEDs knowledge scores of intervention and control groups after education and counseling program? Is there a difference between the daily life activity scores of intervention and control groups after education and counseling program?

Researches offer an education and counseling program about living with CIEDs to patients that having CIEDs for the first time. Participants answers questions in Health Literacy Survey European Questionnaire 16, cardiac implantable electronic devices knowledge scale (researches developed) and Duke Activity Index before education and counseling program, at first month, third month and sixth month after implantation.

Reseraches compare scores between intervention and control groups, also different times in same groups.

ELIGIBILITY:
Inclusion Criteria:

* no communication problems in Turkish
* implanted any type of CIED for the first time
* having low score of HLS EU Q16
* willingness to participate in the study

Exclusion Criteria:

* Not literate
* having vision or hearing problem
* having psychiatric and cognitive impairment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-26 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Baseline knowledge level | Before education
  CIEDs knowledge scale score of patients
Change in knowledge level | At first month after education
  CIEDs knowledge scale score of patients
Change in knowledge level | At third month after education
  CIEDs knowledge scale score of patients
Change in knowledge level | At sixth month after education
  CIEDs knowledge scale score of patients
Baseline daily life activities | Before education
  Duke Activity Index score of patients
Change in daily life activities | At first month after education
  Duke Activity Index score of patients
Change in daily life activities | At third month after education
  Duke Activity Index score of patients
Change in daily life activities | At sixth month after education
  Duke Activity Index score of patients
Baseline health literacy level | Before education
  Health Literacy Survey European Questionnaire 16 score of patients
Change in health literacy level | At first month after education
  Health Literacy Survey European Questionnaire 16 score of patients
Change in health literacy level | At third month after education
  Health Literacy Survey European Questionnaire 16 score of patients
Change in health literacy level | At sixth month after education
  Health Literacy Survey European Questionnaire 16 score of patients

CONTACTS AND LOCATIONS:
Overall Officials: Merve Erünal, Principal Investigator — Dokuz Eylul University Faculty of Nursing; Hatice Mert, Principal Investigator — Dokuz Eylul University Faculty of Nursing
Locations (1):
- Merve Erunal, Balçova, İzmir, Turkey (Türkiye)